CLINICAL TRIAL: NCT03592550
Title: The eValuation of Image Guidance of Stereotactic Body Radiotherapy Using Ultrasound: Assessment in Liver
Acronym: VISUAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4821
Record Dates: First submitted 2018-06-22; First posted 2018-07-19 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group A: Volunteers will be asked to receive ultrasound imaging in repeat voluntary breath hold and during free-breathing.
  Interventions: Device: Ultrasound imaging
- Group B: Volunteers will be asked to receive ultrasound imaging in repeat voluntary breath hold and during free-breathing and in repeat spirometer assisted breath hold.
  Interventions: Device: Ultrasound imaging

INTERVENTIONS:
Device: Ultrasound imaging — Abdominal ultrasound imaging of the liver

SUMMARY:
Worldwide, primary liver cancer is the 3rd most common cause of cancer-related death, accounting for 6% of cancer diagnoses. In the UK, the number of cases reported has more than trebled since the 1970's, with 5550 new cases in 2014 (CRUK statistics 2014). Liver transplant or surgery are the main forms of treatment offered but only less than 20% of patients can tolerate these treatments. There is a need for non-surgical therapies that would improve these patients' chances of survival. Radiotherapy has been shown to increase the likelihood of liver cancer cure. To deliver radiotherapy safely to the patient, the radiation must be delivered to the liver cancer only, avoiding normal liver tissues and other surrounding normal tissues. Because the liver moves during breathing, a liver cancer will also move during radiotherapy. To accurately target the cancer the patient can be asked to hold their breath during treatment to stop the motion. Or motion of the cancer can be monitored and the radiation beam can be moved to follow its motion. The investigators are investigating new methods to either: (a) ensure that when the patient repeats their breath hold the cancer is in the same position each time, or (b) measure the motion of the liver cancer whilst the patient breathes freely. It is not clear which is the best method and therefore are investigating both approaches. Ultrasound is a non-invasive and real-time imaging method that can easily be used to image the liver and may be able to perform both of these tasks. In this study the investigators will test ultrasound equipment, which has been specifically designed to guide radiotherapy. 26 healthy volunteers will be recruited to help evaluate the accuracy of ultrasound to measure the position of the liver in breath hold and in free breathing.

DETAILED DESCRIPTION:
PURPOSE: This observational study of healthy volunteers will test the use of a safe, non-ionising and non-invasive imaging system for the purpose of improving radiotherapy treatment of the liver. This study investigates an image guidance method which may be used to guide liver radiotherapy and enable more accurate treatment on a conventional radiotherapy machine.

RECRUITMENT: Volunteers will need to provide their National Health Service (UK) numbers and be registered on the hospital information system. Volunteers need to be aware that if they are patients at the Royal Marsden Hospital this may raise confidentiality issues. Volunteers will be made aware of this in the recruiting email and the Volunteer Information sheet.

USE OF HEALTHY VOLUNTEERS: This is an observational study, which tests the use of an ultrasound guidance system. The accuracy of the system will be evaluated by comparison of proprietary methods of liver position estimation against a manually derived ground truth derived from the images of the liver acquired in participants. It is not expected that there are any differences in the ultrasound guidance images of healthy volunteers and patients with liver cancer. Ultrasound is a non-invasive and non-ionizing imaging modality with no known side-effects or complications and therefore, safe to use in a volunteer study. Furthermore, this study requires that participants lie on a hard couch for up to 45 minutes and up to 4 times. This would be challenging for the vast majority of patients with liver cancer who are most likely to be frail due to their disease.

REVIEW OF HEALTHY VOLUNTEERS: The ultrasound guidance system provides 3D ultrasound images of the liver for providing positional information only. It is very unlikely that abnormalities will be detectable on 3D US guidance images. These images are not of diagnostic quality, being lower resolution than routine diagnostic 2D ultrasound images. Furthermore, diagnostic ultrasound of the liver often incorporates ultrasound contrast agent, which will not be used in this study. If a radiographer does observe any abnormality, this will be reported to a Consultant Radiologist and the images will be made available for review.

RISKS, BURDENS and BENEFITS: There is very little risk associated with ultrasound and the Automatic Breathing Control (ABC) device, both pieces of the equipment are CE-marked and we are not using outside of their respective intended purposes. The burden to the volunteer is (1) the time spent, (2) the uncomfortable nature of the couch (it has a hard flat surface) and (3) discomfort using the ABC device. The participant will made aware of (1), (2) and (3) by providing details in the volunteer information sheet. Participants who are uncomfortable using the ABC can opt out and still participate in the study. Participants will be able to get up from the couch and walk around to relive any discomfort at any point during the imaging sessions.

There are no benefits for the participants. It is expected that this study will be of benefit to future patients with liver cancer. To ensure there is no perceived benefit of the acquisition of ultrasound images it is stated clearly in the volunteer information sheet that images are not of diagnostic quality and that persons obtaining the images are trained in therapy guidance and not diagnostics, and that images will only be reviewed by a radiologist in the unlikely event that an abnormality is observed.

CONFLICTS OF INTEREST: There are no conflicts of interest. No study investigator will benefit financially from the outcome of this study. The manufacturer of the Clarity ultrasound system will be informed of the results and all results will be published in a peer-reviewed scientific journal.

ACCESS to DATA: The investigators wish to make anonymised image data available to other researchers on request for the purpose of medical research. This is intended to maximise the value of the data and may provide greater benefit to patients. Volunteers will be asked to consent to their anonymised data being made available to other researchers.

AIMS: This study aims to develop and evaluate the use of 3 ultrasound (3DUS) to estimate the liver position for radiotherapy guidance. This is an exploratory study, where Clarity US of the abdomen will be acquired in healthy volunteers. 3D US-sim, 3D US-guide, 3D US-monitor and 4D US-monitor will be used to meet the following study objectives:

1. The accuracy of B-mode 3D US-guide, to estimate the position of the liver in breath-hold for verification of (1) daily set-up position (set-up US-guide) and (2) repeat breath hold relevant to radiotherapy delivery (BH 3D US-monitor), will be determined. Accuracy will be assessed by comparison of US-guide and US-monitor determined liver position with a manually determined 'gold standard' liver position.
2. Comparison of the accuracy of power Doppler and B-mode US-guide/US-monitor for the estimation of liver position during breath hold.
3. Assessment of the accuracy of 4D US-monitor to estimate liver motion during free breathing (FB).
4. Comparison of liver position stability using spirometry and voluntary breath-hold (vBH) using US-monitoring.
5. Assessment of the availability of a second or third ultrasound field of view for increasing the accuracy of US-guide based estimates of liver motion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers.

Exclusion Criteria:

* Healthy volunteers who are unable to hold their breath for 30 seconds in exhalation.
* Healthy volunteers who are unable to lie for extended period of time (up to 45 minutes including short breaks of a few minutes) on a hard surface (treatment couch).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers drawn from staff at ICR and Royal Marsden Hospital
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Difference in liver position after set-up | Within 2 months of image acquisition
  The mean difference in liver position measured by US-guide and using the gold standard method, measured in millimetres in the superior-inferior (SI), anterior-posterior (AP) and left-right (LR) directions over 5 set-up sessions.

SECONDARY OUTCOMES:
Difference in liver position during repeat breath hold | Within 2 months of image acquisition
  The mean difference in liver position measured by US-guide and using the gold standard method, measured in millimetres in the superior-inferior (SI), anterior-posterior (AP) and left-right (LR) directions over 3 breath holds.
Difference in liver position after set-up using Doppler ultrasound and US-guide | Within 2 months of image acquisition
  The mean difference in liver position measured by B-mode US-guide and using the Doppler US-guide method, measured in millimetres in the superior-inferior (SI), anterior-posterior (AP) and left-right (LR) directions over 5 set-ups.
Liver position during free-breathing | Within 2 months of image acquisition
  The liver position measured in the SI, AP and LR directions, measured by 4D US-monitor during free breathing.
Liver motion between fractions and repeat thresholds | Within 2 months of image acquisition
  The mean motion of the liver during voluntary breath-hold and assisted breath-hold measured using the gold standard method.
Number of available imaging positions | Within 2 months of image acquisition
  The number of imaging positions (1 2 or 3), which may be used by 4D US-guide to accurately measure liver position during free-breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Harris, PhD, Principal Investigator — Institute of Cancer Research, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data will be available on request